CLINICAL TRIAL: NCT03812549
Title: Multi-center Phase I Study of Sintilimab in Combination With Radiotherapy in Treatment Naive PD-L1 Positive Stage IV Non-small Cell Lung Cancer (NSCLC)
Brief Title: Safety and Tolerability Evaluation of Sintilimab in Combination With Radiation in Stage IV NSCLC Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, You Lu, Chair of Department of Thoracic Oncology, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHC-001
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Stage IV NSCLC
Keywords: Immunotherapy;SBRT; PD-L1 positive; LDRT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; Radiosurgery; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab Combined with SBRT and LDRT (Experimental): Period 1-Dose escalation cohort. Dose Level 1: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT, 2 Gy in 1 fraction) + anti-PD-1 inhibitor 200mg.
  Dose Level 2: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT, 4 Gy in 2 fractions) + anti-PD-1 inhibitor 200mg.
  Dose Level 3: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT, 10 Gy in 5 fractions) + anti-PD-1 inhibitor 200mg.
  Period 2 - Expansion cohort. SBRT dose at 30 Gy/3f + LDRT + anti-PD-1 inhibitor 200mg, LDRT dose at RDE determined in Period 1.
  Interventions: Drug: Sintilimab; Radiation: stereotactic body radiation therapy; Radiation: Low Dose Radiotherapy

INTERVENTIONS:
Drug: Sintilimab — Patients will receive treatment with Sintilimab 200mg every 3 weeks for a maximum of 24 months.
  Other Names: IBI308
Radiation: stereotactic body radiation therapy — Radiation treatment utilized in this trial consists of SBRT with a standard doses to 30 Gy/3f
  Other Names: SBRT
Radiation: Low Dose Radiotherapy — LDRT at dose escalation levels: 2 Gy/1f, 4 Gy/2f, 10 Gy/5f with conventional external beam radiation.
  Other Names: LDRT

SUMMARY:
This pilot phase I trial aims to investigate the safety and tolerability of anti-programmed cell death-1 (PD-1) monoclonal antibody Sintilimab (also called IBI308) in combination with concurrent stereotactic body radiation therapy (SBRT) and low dose radiotherapy (LDRT) in treating patients with stage IV non-small cell lung cancer (NSCLC).

At least 29 participants will be enrolled in this study. All will take part at West China Hospital, Sichuan University.

DETAILED DESCRIPTION:
This exploratory phase I study will be conducted in two steps:

Step A: A low dose radiotherapy (LDRT) dose escalation, 6 patients per cohort (a total of 18 patients) will be enrolled to determine the maximum tolerated dose (MTD), dose-limiting toxicity (DLT) and recommended dose for expansion (RDE) for lung LDRT.

Step B: A lung LDRT dose expansion

All eligible patients will receive lung SBRT dosed at 30 Gy in 3 fractions, in combination with LDRT at different dose levels (decried as below) starting from the 2nd day of SBRT, followed by sintilimab monotherapy starting within 7 days after radiation completed. Sintilimab will be given at 200mg every 3 weeks until disease progression, unacceptable toxicities, the patient withdraws informed consent, or sintilimab reaches a maximum of up to 24 months.

Patients in the dose escalation will receive lung LDRT at 3 cohorts with increasing dose levels: 2 Gy in 1 fraction in dose level 1, 4 Gy in 2 fractions in dose level 2, 10Gy in 5 fractions in dose level 3.

A cohort of 17 patients will receive lung LDRT at the RDE determined during the dose escalation phase in combination with SBRT and Sintilimab to obtain additional safety and response data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed stage IV NSCLC.
2. Enough tumor tissue samples.
3. No previous radiation, chemotherapy, immunotherapy. Patients who have received neoadjuvant or adjuvant chemotherapy 12 months before enrollment is permitted.
4. At least three measurable disease according to RECIST 1.1 that meet SBRT and LDRT radiation requirement as protocol defined
5. PD-L1 expression positive (TPS >1%)
6. Be ≥18 years of age on day of signing informed consent and ≤75 years old.
7. ECOG 0-1.
8. Patients must have normal organ and marrow function as defined below: Total bilirubin </= 1.5 mg/dL. Aminotransferase (AST) Serum Glutamic Oxaloacetic Transaminase (SGOT)/ Alanine Aminotransferase (ALT) Serum Glutamic-Pyruvic Transaminase (SGPT) <2.5 X institutional upper limit of normal (patients with liver involvement will be allowed </= 5.0 X institutional upper normal limit) *WBC >/= 3500/uL, ANC >/= 1500/uL *Platelets >/= 90K *Hemoglobin >/= 9g/dL *Creatinine </= 1.5 x ULN.
9. Be willing and able to provide written informed consent/assent for the trial.
10. Patients should be able to tolerate a course of radiotherapy as assessed by the investigator.
11. No contradiction to radiation per radio-oncologists' judgments
12. Life expectancy of > 6 months.

Exclusion Criteria:

1. EGFR/ALK/ROS-1 mutation or mutation status unknown.
2. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
3. Subjects with coronary bypass operation.
4. Subjects with insufficient heart function, liver function and kidney function.
5. Subjects with severe uncontrollable psychotic symptoms.
6. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, anti-tumor necrosis factor agents) within 4 weeks prior to enrollment or anticipated requirement for systemic immunosuppressive medications during the trial.
7. Subjects with active, known or suspected autoimmune disease such as interstitial pneumonia, uveitis, Crohn's disease, autoimmune thyroiditis. Subjects with cured childhood asthma, type I diabetes mellitus only requiring hormone replacement.
8. Known history of allogeneic organ or allogeneic hemopoietic stem cell transplantation.
9. Known hypersensitivity or allergy to monoclonal antibody.
10. Subjects with a history of interstitial lung disease.
11. Uncontrolled concomitant disease, including but not limited to :

1)Active or poorly controlled severe infection 2)Human Immunodeficiency Virus (HIV) infection (HIV antibody positive) 3)Known acute or chronic active hepatitis B (HBV DNA positive) infection or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive) infection 4)Active tuberculosis 5)Symptomatic congestive heart failure (New York Heart Association grade III-IV) or symptomatic, poorly controlled arrhythmia 6)Uncontrolled hypertension (SBP ≥ 160mmHg or DBP ≥ 100mmHg) 7)Prior arterial thromboembolism event, including myocardial infarction, unstable angina, stroke and transient ischemic attack, within 6 months of enrollment 8)Concomitant disease needs anticoagulant therapy 9)Uncontrolled hypercalcemia（Ca2+>1.5mmol/L or Ca >12mg/dl or corrected Serum Calcium >ULN），or Symptomatic hypercalcemia during diphosphonate therapy

12. Other primary malignancy, with the exception of: (radical Non-melanoma skin cancer or cured cervical in-situ carcinoma;).

13. Subjects with other diseases or abnormal Lab test results which might increase the risk of enrollment and treatment or Interfere with the interpretation of study results could be excluded according to the judgments of investigator.

14. Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma P, Allison JP. The future of immune checkpoint therapy. Science. 2015 Apr 3;348(6230):56-61. doi: 10.1126/science.aaa8172. PMID 25838373
- [Background] Demaria S, Coleman CN, Formenti SC. Radiotherapy: Changing the Game in Immunotherapy. Trends Cancer. 2016 Jun;2(6):286-294. doi: 10.1016/j.trecan.2016.05.002. PMID 27774519
- [Background] Kaur P, Asea A. Radiation-induced effects and the immune system in cancer. Front Oncol. 2012 Dec 17;2:191. doi: 10.3389/fonc.2012.00191. eCollection 2012. PMID 23251903
- [Background] Bernstein MB, Krishnan S, Hodge JW, Chang JY. Immunotherapy and stereotactic ablative radiotherapy (ISABR): a curative approach? Nat Rev Clin Oncol. 2016 Aug;13(8):516-24. doi: 10.1038/nrclinonc.2016.30. Epub 2016 Mar 8. PMID 26951040
- [Background] Park SS, Dong H, Liu X, Harrington SM, Krco CJ, Grams MP, Mansfield AS, Furutani KM, Olivier KR, Kwon ED. PD-1 Restrains Radiotherapy-Induced Abscopal Effect. Cancer Immunol Res. 2015 Jun;3(6):610-9. doi: 10.1158/2326-6066.CIR-14-0138. Epub 2015 Feb 19. PMID 25701325
- [Background] Postow MA, Callahan MK, Barker CA, Yamada Y, Yuan J, Kitano S, Mu Z, Rasalan T, Adamow M, Ritter E, Sedrak C, Jungbluth AA, Chua R, Yang AS, Roman RA, Rosner S, Benson B, Allison JP, Lesokhin AM, Gnjatic S, Wolchok JD. Immunologic correlates of the abscopal effect in a patient with melanoma. N Engl J Med. 2012 Mar 8;366(10):925-31. doi: 10.1056/NEJMoa1112824. PMID 22397654
- [Background] Du J, Su S, Li H, Shao J, Meng F, Yang M, Qian H, Zou Z, Qian X, Liu B. Low dose irradiation increases adoptive cytotoxic T lymphocyte migration in gastric cancer. Exp Ther Med. 2017 Dec;14(6):5711-5716. doi: 10.3892/etm.2017.5305. Epub 2017 Oct 13. PMID 29285113
- [Background] Brooks ED, Chang JY. Time to abandon single-site irradiation for inducing abscopal effects. Nat Rev Clin Oncol. 2019 Feb;16(2):123-135. doi: 10.1038/s41571-018-0119-7. PMID 30401936

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 2Gy in 1 Fraction: DOSE LEVEL 1: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT, 2Gy/1f) + anti-PD-1 inhibitor 200mg.
- Dose Level 2: 4Gy in 2 Fractions: DOSE LEVEL 2: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT, 4Gy/2f) + anti-PD-1 inhibitor 200mg.
- Dose Level 3: 10Gy in 5 Fractions: DOSE LEVEL 3: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT, 10Gy/5f) + anti-PD-1 inhibitor 200mg.
Period: Dose Level 1: 2Gy in 1 Fraction
Arm/Group | Dose Level 1: 2Gy in 1 Fraction | Dose Level 2: 4Gy in 2 Fractions | Dose Level 3: 10Gy in 5 Fractions
Started | 6 | 0 | 0
Completed | 6 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Dose Level 2: 4Gy in 2 Fractions
Arm/Group | Dose Level 1: 2Gy in 1 Fraction | Dose Level 2: 4Gy in 2 Fractions | Dose Level 3: 10Gy in 5 Fractions
Started | 0 | 17 | 0
Completed | 0 | 17 | 0
Not Completed | 0 | 0 | 0
Period: Dose Level 3: 10Gy in 5 Fractions
Arm/Group | Dose Level 1: 2Gy in 1 Fraction | Dose Level 2: 4Gy in 2 Fractions | Dose Level 3: 10Gy in 5 Fractions
Started | 0 | 0 | 6
Completed | 0 | 0 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: 2Gy in 1 Fraction | Dose Level 2: 4Gy in 2 Fractions | Dose Level 3: 10Gy in 5 Fractions | Total
Number analyzed (Participants) | 6 | 17 | 6 | 29
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.3 [52.2 to 71.5] | 68.2 [47.2 to 74.8] | 64.3 [50.1 to 68.5] | 65.0 [47.2 to 74.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3
  Male | 5 | 15 | 6 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 17 | 6 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 6 | 17 | 6 | 29
smoking history [Number; unit: participants] | 5 | 15 | 4 | 24
PD-L1 expression ≥ 50% [Number; unit: participants] | 2 | 7 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and/or Dose Limiting Toxicities of Sintilimab in Combination With SBRT and LDRT
Description: Adverse Events and/or Dose Limiting Toxicity graded per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Time Frame: from randomization through 30 days after last dosing, up to 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: 2Gy in 1 Fraction: DOSE LEVEL: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT) dose from 2 Gy to 10Gy + anti-PD-1 inhibitor 200mg.
  Therefore, there were 3 different dose levels.
  DOSE LEVEL 1: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT, 2Gy/1f) + anti-PD-1 inhibitor 200mg.
- Dose Level 3: 10Gy in 5 Fractions: DOSE LEVEL 1: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT, 10Gy/5f) + anti-PD-1 inhibitor 200mg.
Arm/Group | Dose Level 1: 2Gy in 1 Fraction | Dose Level 2: 4Gy in 2 Fractions | Dose Level 3: 10Gy in 5 Fractions
Number analyzed (Participants) | 6 | 17 | 6
Participants
  Any TRAE Grade ≥ 3 | 0 | 5 | 1
  Any TRAE Grade < 3 | 6 | 12 | 5

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Investigator assessed PFS according to RECIST v1.1. Progression free survival is defined as time of enrollment to first evidence of progressive disease.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: up to 24 months after the enrollment
Measure: Median (95% Confidence Interval); unit: month
Groups:
- Dose Level 3: 10Gy in 5 Fraction: DOSE LEVEL 3: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT, 10Gy/5f) + anti-PD-1 inhibitor 200mg.
Arm/Group | Dose Level 1: 2Gy in 1 Fraction | Dose Level 2: 4Gy in 2 Fractions | Dose Level 3: 10Gy in 5 Fraction
Number analyzed (Participants) | 6 | 17 | 6
month | 7.228 [0 to 17.323] | 9.035 [1.122 to 16.948] | 4.501 [0 to 12.861]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Investigator assessed ORR using RECIST v1.1 including the all tumor, the tumor undergoing LDRT and the tumor which do not receive radiotherapy.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: up to 24 months after the enrollment
Population: objective response rate
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 2: 4Gy in 2 Fraction: DOSE LEVEL 2: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT, 4Gy/2f) + anti-PD-1 inhibitor 200mg.
Arm/Group | Dose Level 1: 2Gy in 1 Fraction | Dose Level 2: 4Gy in 2 Fraction | Dose Level 3: 10Gy in 5 Fraction
Number analyzed (Participants) | 6 | 16 | 6
Participants | 4 | 10 | 3

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the difference (in months) between the date of study enrollment to the date death due to any cause
Time Frame: up to 24 months after the enrollment
Population: overall survival
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Dose Level 1: 2Gy in 1 Fraction | Dose Level 2: 4Gy in 2 Fractions | Dose Level 3: 10Gy in 5 Fractions
Number analyzed (Participants) | 6 | 17 | 6
years | NA [NA to NA] — insufficient number of participants with events | NA [NA to NA] — insufficient number of participants with events | 15.639 [0 to 32.8]

ADVERSE EVENTS:
Time Frame: from randomization through 30 days after last dosing，up to 24 months
Description: Adverse events (AEs) were monitored during the study and summarized according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
Groups:
- Dose Level 1: Dose level 1: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT) dose at 2Gy/1f + anti-PD-1 inhibitor 200mg.
- Dose Level 2: Dose level 2: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT) dose at 4Gy/2f + anti-PD-1 inhibitor 200mg.
- Dose Level 3: Dose level 3: Stereotactic body radiation therapy (SBRT) dose at 30 Gy/3f + Low Dose Radiotherapy (LDRT) dose at 10Gy/5f + anti-PD-1 inhibitor 200mg.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/17 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 5/17 | 1/6
Other Adverse Events (participants affected / at risk) | 6/6 | 12/17 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=17) | Dose Level 3 (N=6)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylaxis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoadrenocorticism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=17) | Dose Level 3 (N=6)
Hypothyroidism (Endocrine disorders) | 3 (3) | 6 (6) | 1 (1)
ALT increased (Hepatobiliary disorders) | 3 (3) | 5 (5) | 1 (1)
AST increased (Hepatobiliary disorders) | 2 (2) | 4 (4) | 3 (3)
Hypoproteinemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 2 (2)
Cardiac arrhythmia (Cardiac disorders) | 0 (0) | 4 (4) | 2 (2)
Fatigue (General disorders) | 0 (0) | 3 (3) | 2 (2)
ACTH increased (Endocrine disorders) | 2 (2) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT03812549/Prot_SAP_000.pdf